CLINICAL TRIAL: NCT02483247
Title: A Phase Ib/II Clinical Study of BBI503 in Combination With Selected Anti-Cancer Therapeutics in Adult Patients With Advanced Cancer
Brief Title: A Study of BBI503 in Combination With Selected Anti-Cancer Therapeutics in Adult Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBI503-201
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Cancer
Keywords: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Capecitabine; Doxorubicin; liposomal doxorubicin; Nivolumab; pembrolizumab; Paclitaxel; Sunitinib

ARMS (6):
- Combo with Capecitabine (Experimental)
  Interventions: Drug: BBI503; Drug: Capecitabine
- Combo with Doxorubicin (Experimental)
  Interventions: Drug: BBI503; Drug: Doxorubicin
- Combo with Nivolumab (US only) (Experimental)
  Interventions: Drug: BBI503; Drug: Nivolumab
- Combo with Pembrolizumab (Experimental)
  Interventions: Drug: BBI503; Drug: Pembrolizumab
- Combo with Paclitaxel (Experimental)
  Interventions: Drug: BBI503; Drug: Paclitaxel
- Combo with Sunitinib (Experimental)
  Interventions: Drug: BBI503; Drug: Sunitinib

INTERVENTIONS:
Drug: BBI503 — Patients in this trial will receive BBI503 orally, daily, and continuously. The dose-level of BBI503 will be assigned according to the dose-cohort open at the time the patient enrolls into a given arm. The study-arm and combination anti-cancer agent for a given patient will be determined by the investigator. BBI503 Dose Level 1: 200 mg once daily, Dose Level 2: 300 mg once daily.
  Other Names: amcasertib; BBI-503; BB503
Drug: Capecitabine — Capecitabine 1000 mg/m^2 body surface area is administered orally, twice daily, on days 1-14 of each 21 day cycle.
  Other Names: Xeloda
  Arms: Combo with Capecitabine
Drug: Doxorubicin — Doxorubicin 60 mg/m^2 body surface area is administered intravenously once every three weeks (21-days).
  Other Names: Doxil; Adriamycin
  Arms: Combo with Doxorubicin
Drug: Nivolumab — Nivolumab 3 mg/kg is administered as an intravenous infusion over 60 minutes on day 1 and day 15 of each 28 day cycle.
  Other Names: Opdivo
  Arms: Combo with Nivolumab (US only)
Drug: Pembrolizumab — Pembrolizumab 2 mg/kg is administered as an intravenous infusion over 30 minutes once every three weeks (21-days).
  Other Names: Keytruda
  Arms: Combo with Pembrolizumab
Drug: Paclitaxel — Paclitaxel 80 mg/m^2 body surface area is administered intravenously once weekly on day 1, day 8, and day 15 of each 28 day cycle.
  Other Names: Taxol
  Arms: Combo with Paclitaxel
Drug: Sunitinib — Sunitinib 37.5 mg is administered once daily.
  Other Names: Sutent
  Arms: Combo with Sunitinib

SUMMARY:
This is an open label, multi-center, Phase 1/2 study of BBI503 administered in combination with selected anti-cancer therapeutics in adult patients with advanced cancer. The goal of the study is to determine the safety, tolerability, and RP2D of BBI503 in combination with each of the selected anti-cancer agents.

ELIGIBILITY:
Major inclusion criteria:

1. A histologically or cytologically confirmed solid tumor that is locally advanced, recurrent, or metastatic; for which curative resection is not currently possible; and for which systemic treatment with one of the selected anti-cancer agents is a reasonable therapeutic option.
2. Must be ≥ 18 years of age
3. Has disease such that progression or response to therapy can be evaluated objectively while on protocol.
4. Must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Male or female patients of childbearing potential must agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after the last dose.
6. Females of childbearing potential must have a negative serum pregnancy test.
7. Must have aspartate transaminase (AST) ≤ 2.5 × upper limit of normal (ULN) and alanine transaminase (ALT) ≤ 2.5 × ULN. Patients who do not have hepatocellular carcinoma but who have liver lesions or liver metastases may be eligible if AST ≤ 3.5 × ULN and AST ≤ 3.5 × ULN if agreed upon by the investigator and medical monitor for the sponsor.
8. Hemoglobin (Hgb) ≥ 9 g/dl
9. Total bilirubin ≤ 1.5 × ULN. For patients with liver lesions, total bilirubin ≤ 2.0 × ULN may be enrolled if agreed upon by the investigator and medical monitor for the sponsor
10. Creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional upper limit of normal (using the Cockcroft-Gault equation).
11. Absolute neutrophil count ≥ 1.5 × 10^9/L
12. Platelets ≥ 100 × 10^9/L
13. Life expectancy ≥ 3 months

Major exclusion criteria:

1. Received anti-cancer chemotherapy, radiotherapy, immunotherapy, or investigational agents within 7 days of first dose of protocol therapy. Patients may begin protocol therapy on a date determined by the investigator and medical monitor for the sponsor after a minimum of 7 days since last receiving anti-cancer treatment, provided that all adverse events related to that have resolved or have been deemed irreversible.
2. Major surgery within 4 weeks prior to first dose; major surgery is defined as a procedure requiring any of the following: general anesthesia, intubation and mechanical ventilation, or major incision (e.g., thoracotomy, laparotomy)
3. Any known, untreated, brain metastases. Patients with treated brain metastases must have no clinical symptoms from the metastases, and must be either off steroids or on a stable dose of steroids ≤ 10 mg prednisone or equivalent for at least 2 weeks prior to protocol enrollment. Patients with known leptomeningeal metastases are excluded, even if treated.
4. Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study.
5. Significant gastrointestinal disorder(s), in the opinion of the Principal Investigator, such as active inflammatory bowel disease, extensive gastric or small intestinal resection (which has resulted in short-gut syndrome or the inability to take oral medications).
6. Unable or unwilling to swallow either BBI503 daily or an oral selected anti-cancer therapeutics; or, unwilling to receive intravenous injection of IV anti-cancer therapeutics.
7. Positive for Human Immunodeficiency Virus (HIV), Hepatitis B (Hepatitis B Surface Antigen [HBsAg] reactive), or Hepatitis C virus (Hepatitis C Virus Ribonucleic Acid (HCV RNA] (qualitative) is detected).
8. Uncontrolled concurrent illness including, but not limited to: ongoing or active infection requiring therapy, clinically significant non-healing or healing wounds, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or on mild exertion), uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements
9. Subjects with a history of another primary cancer with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; c) localized prostate cancer not requiring systematic therapy; and d) other primary cancer with no known active disease present, and no treatment administered in the 2 years prior to enrollment.
10. For patients to be treated with a regimen containing capecitabine: a) Known hypersensitivity to capecitabine, b) Known dihydropyrimidine dehydrogenase (DPD) deficiency, c) Significant gastrointestinal disorder(s) that would, in the opinion of the Investigator, prevent absorption of an orally available agent
11. For patients to be treated with a regimen containing sunitinib: a) Uncontrolled hypertension (systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management), b) Evidence of bleeding diathesis or a clinically significant coagulopathy (≥ CTCAE Grade 3) within 4 weeks prior to the start of study, c) Recent hypoglycemia, d) Uncontrolled thyroid dysfunction despite optimal medical therapy
12. For patients to be treated with a regimen containing doxorubicin: a) Known left ventricular ejection fraction < 50%, b) Hypersensitivity to doxorubicin
13. A patient to be treated with a regimen containing nivolumab or pembrolizumab will be excluded if the patient: a) Has an active autoimmune disease requiring immunosuppression with the exception of subjects with isolated vitiligo, resolved childhood asthma or atopic dermatitis, controlled hypoadrenalism or hypopituitarism, and euthyroid patients with a history of Grave's disease, b) Has had a previous life-threatening (CTCAE grade 4) immune-mediated adverse reaction; or, a previous severe (CTCAE grade 3) immune mediated adverse reaction that required treatment with corticosteroids (more than 10 mg/day prednisone or equivalent dose) for longer than 12 weeks, c) Has a transplanted organ, d) Has interstitial lung disease or active, non-infectious pneumonitis, e) Has received a live vaccine within 30 days prior to first dose, f) Previous severe hypersensitivity reaction to another monoclonal antibody (mAb), g) Has been treated with another monoclonal antibody ≤ 4 weeks before first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2015-09; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Determination of the safety and tolerability of BBI503 administered in combination with selected anti-cancer therapeutics by assessing dose-limiting toxicities (DLTs) | 3 or 4 weeks based on the cycle of the selected anti-cancer therapeutics
Determination of the Recommended Phase 2 Dose (RP2D) by assessing dose-limiting toxicities (DLTs) | 3 or 4 weeks based on the cycle of the selected anti-cancer therapeutics

SECONDARY OUTCOMES:
Assessment of the preliminary anti-tumor activity by performing tumor assessments every 8 weeks (Phase 2 portion) | 6 months
  Evaluation of anti-tumor activity will be performed according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Pharmacokinetic profile of BBI503 administered in combination with selected anti-cancer therapeutics as assessed by maximum plasma concentration and area under the curve | 0, 1, 2, 3, 4, 6, 8, 10, 24 hours on day 1, cycles 1 and 2
Pharmacodynamic activity of BBI503 administered in combination with selected anti-cancer therapeutics as assessed by biomarker analysis | 3 or 4 weeks based on the cycle of the selected anti-cancer therapeutics
  Histopathology and Cancer Stem Cell assays will be performed to provide information of the biomarkers on biopsied patient tumor tissue, and archival samples.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - Parkview Research Center, Fort Wayne, Indiana
  - Indiana University Health Goshen, Goshen, Indiana
  - Indiana University -Ball, Indianapolis, Indiana
  - Indiana University-SCC, Indianapolis, Indiana
  - Louisiana State Univesity, New Orleans, Louisiana
  - US Oncology Research, Fairfax, Virginia
- Canada (2):
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario